CLINICAL TRIAL: NCT05040282
Title: The Rate and Predictors of Amenorrhea at 1-year Follow-up in Women Using Etonogestrel Implant
Brief Title: The Amenorrhea With Etonogestrel Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant professor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Implanon-nxt
Record Dates: First submitted 2021-08-21; First posted 2021-09-10 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Etonogestrel 68 mg implant (Other): Women will be subjected to etonogestrel 68 mg implant insertion (Implanon NXT; Organon, USA Inc) according to manufacture instructions. The insertion will be within the first 5 days of the menstrual cycle
  Interventions: Device: Implanon NXT

INTERVENTIONS:
Device: Implanon NXT — women will be subjected to etonogestrel 68 mg implant insertion. Participants will be trained on how to fill the menstrual diary. The menstrual diary includes information about days of bleeding and spotting days.
  Other Names: Etonogestrel subdermal implant

SUMMARY:
The etonogestrel subdermal implant has been available worldwide for more than 15 years. The action of etonogestrel subdermal implant is principal via suppression of ovulation, but it also has effects on cervical mucus and in some women induces suppression of endometrial proliferation. Several studies have confirmed its high efficacy and convenience. The uterine bleeding problems and in particular irregular bleeding and amenorrhea are major side effects of etonogestrel subdermal implant. A considerable number of patients request early removal due to bleeding changes. Amenorrhea occurs in about 22% in etonogestrel subdermal implant users. Despite the presence of many studies that reported the prevalence of etonogestrel subdermal implant-associated bleeding, little is known about the predictive factors affecting menstrual bleeding patterns especially amenorrhea after etonogestrel subdermal implant insertion. These predictive factors should be provided prior to the etonogestrel subdermal implant insertion which may improve acceptance and continuation of etonogestrel subdermal implant.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 18 and 40 years.
2. Women who are not lactating.
3. Non-pregnant women
4. Women have regular menstrual cycles every 21-35 days with a typical cycle length variation of no more than 5 days.
5. Women who will ESI only for pregnancy prevention for at least 12 months.
6. Have not any medical or gynecologic problems.

Exclusion Criteria:

1. Women with any contraindications for progesterone-only contraception in accordance with WHO eligibility criteria.
2. Refuse participation in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Number of women with amenorrhea after using etonogestrel subdermal implant | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided